CLINICAL TRIAL: NCT04609956
Title: Comparative Randomized Study of Virtual Reality Technology on Pain Perception and Anxiety Levels in Adolescents and Young Adults During Third Molar Germ Avulsion Surgery
Brief Title: Virtual Reality Technology on Pain Perception and Anxiety Levels in Adolescents and Young Adults During Third Molar Germ Avulsion Surgery (VIDAMO)
Acronym: VIDAMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 29BRC20.0107
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anxiety, Dental
Keywords: virtual reality; oral surgery; anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study is a monocentric interventional prospective comparative randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality (Experimental): Experimental arm is a virtual reality headphones
  Interventions: Other: Virtual reality
- standard (Other): Control arm is a usual practice (hydroxyzine + patient music with headphones)
  Interventions: Other: Standard

INTERVENTIONS:
Other: Virtual reality — Virtual reality consists of a headphones, a virtual reality headset and a smartphone.
  Arms: virtual reality
Other: Standard — Standard arm is the habitual procedure. They use hydroxyzine and music with headphones
  Arms: standard

SUMMARY:
For a long time, the fear of the dental surgeon has been the main reason why a percentage of the population avoids regular consultation.

There are many techniques to manage anxiety (tell-show-do, positive reinforcement, live modeling, etc). Now, virtual reality offers this possibility as a non-drug alternative technique.

Few studies have assessed the value of virtual reality in peroperative during an oral surgery procedure.

It is interesting to compare the immediate post-operative anxiety level between groups using virtual reality headset (RV) versus standard protocol (hydroxyzine + music with headphones : SMP)

DETAILED DESCRIPTION:
Anxiety is defined as a state of psychic disorder caused by fear of danger ; pain as an unpleasant sensory and emotional experience. Although pain and anxiety are subjective sensations, oral cavity care is very much associated with these perceptions.

Thus, the fear of the oral health practitioner (dental surgeon, oral surgeon, maxillofacial surgeon, etc.) is one of the main reasons why a large part of the population does not consult. This real phobia installed in people's imaginary is partly explained by the fact that the mouth is an intimate part of the body. Indeed, according to the Freudian theory, discovery of body and sexuality begins with the oral stage with the oral and esophageal sphere favored as an erogenous zone (supported by the motor activity of sucking). In this way, the oral cavity is a place of love privacy and erotic intimacy, but also a means of communication and a means of recognizing tastes. Regular consultation with a specialist is consequently essential since good oral hygiene is a source of well-being (notions of pleasure, satisfaction).

Oral health practitioners have many solutions in order to reduce patients' apprehension of anxiety and their painful perceptions. In addition to the psychological approach and cognitive-behavioral therapy (tell-show-do, adapt vocabulary, involve the patient in the therapeutic project) ; medical means are available to the practitioner. According to the therapeutic gradient: firstly use of anxiolytics (hydroxyzine) more or less associated with music therapy or other methods of distraction, conscious sedation (Equimolar mixture of Oxygen and Nitrous Oxide - EMONO) and as a last resort general anesthesia.

An alternative non-drug technique has increased : the use of virtual reality (VR). This new technology, recognized for its entertainment value (creation of virtual environments that immerse people in a simulated world) has been extended to other fields including health, particularly for pain and anxiety management.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 14 and 20 years
* Needing one (or more) germ avulsion (s) of the third molars
* With asymptomatic tooth, no signs of infection and germ status
* Affiliated or beneficiary of a social security system
* Have given informed consent or whose consent has been given by one parent

Exclusion Criteria:

* Patients with visual or auditory deficits that contra-indicating the use of the virtual reality headset
* Non-cooperative patients, who do not speak or do not read French fluently, don't understand the principle of a stress scale and collaborate on tests.
* Refusal to participate

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-16 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Modified Anxiety Dental Scale (MADS) | Day 0
  For primary outcome, (Modified anxiety dental scale (MADS) is a questionnaire measuring immediate post-operative anxiety. MADS is assessed on a 0 (no stressed) to 25 (very stressed) scale. A score greater than 19 or more corresponds to a very stressed or even phobic patient.

SECONDARY OUTCOMES:
Modified Anxiety Dental Scale (MADS) | Day 0
  For second outcome, (Modified anxiety dental scale (MADS) is a questionnaire measuring pre-operative anxiety. MADS is assessed on a 0 (no stressed) to 25 (very stressed) scale. A score greater than 19 or more corresponds to a very stressed or even phobic patient.
Modified Anxiety Dental Scale (MADS) | Day 7
  For second outcome, (Modified anxiety dental scale (MADS) is a questionnaire measuring delay post-operative anxiety.MADS is assessed on a 0 (no stressed) to 25 (very stressed) scale. A score greater than 19 or more corresponds to a very stressed or even phobic patient.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, Finistère, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest University Hospital. Requestors will be required to sign and complete a data access agreement.